CLINICAL TRIAL: NCT00013208
Title: Proactive Diabetes Case Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIR 97-077
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Case Management

INTERVENTIONS:
Behavioral: Case Management

SUMMARY:
Despite a growing array of therapeutic options and efficacious treatment strategies to prevent or delay some of the most severe complications of type 2 diabetes, there continue to be many individuals with outcomes that are far from optimal. Interventions to improve diabetes care by educating providers and patients have been disappointing. In the past several years, case management has been widely advocated as a cost-effective approach to coordinate diabetes care and improve outcomes, although there is little rigorous evidence demonstrating the benefits of this type of intervention.

DETAILED DESCRIPTION:
Background:

Despite a growing array of therapeutic options and efficacious treatment strategies to prevent or delay some of the most severe complications of type 2 diabetes, there continue to be many individuals with outcomes that are far from optimal. Interventions to improve diabetes care by educating providers and patients have been disappointing. In the past several years, case management has been widely advocated as a cost-effective approach to coordinate diabetes care and improve outcomes, although there is little rigorous evidence demonstrating the benefits of this type of intervention.

Objectives:

This study had the following specific aims: 1) to evaluate the effect of a targeted, proactive case management intervention for high risk veterans with type 2 diabetes on: a) glycemic control, b) intermediate cardiovascular outcomes, c) satisfaction, d) adherence to specific care standards, and e) short-term resource utilization; and 2) using Monte Carlo simulation models, to estimate the expected impact of changes in key processes of care and intermediate outcomes on end-stage outcomes.

Methods:

This study was conducted as a prospective randomized controlled trial. Participating veterans with diabetes (N = 246) receiving care at two VAMCs were randomly assigned, stratified by site and baseline hemoglobin A1c (A1c), to the intervention or control group. The intervention consisted of two nurse practitioners who actively monitored and coordinated patient care, guided by approved treatment algorithms. Data for the study were collected through a baseline and exit examination, a baseline and exit survey, and the VA medical information system. The primary outcome measure was the change in glycemic control, as measured by A1c. Secondary outcomes included serum LDL, blood pressure, satisfaction, and resource utilization. The data were analyzed using univariate and bi-variate (t-test, Wilcoxon rank-sum, chi-square) methods as well as multivariable regression.

Status:

Completed Manuscripts

ELIGIBILITY:
Inclusion Criteria:

Patients were eligible to participate in the study if their most current hemoglobin A1c (HbA1c) was >=8.5 (reported within the last year); they had at least 1 prescription for an oral hypoglycemic agent, insulin, or monitoring supplies filled in the last year; and, they had an outpatient visit scheduled with a general internist, nurse practitioner, or physician assistant between May, 1999 and January, 2000.

Patients were not eligible for the study if the patient (or another member of the household when applicable) indicated that they: (1) were under 18 years of age; (2) had never been diagnosed with diabetes; (3) had been diagnosed with Type 1 diabetes or had been diagnosed before age 30; (4) did not have a telephone; (5) did not speak English; (6) were not competent for interview; (7) did not receive their primary diabetes care within the VA system; (8) were currently receiving treatment for cancer (other than non-melanoma); (9) had been diagnosed with kidney failure, congestive heart failure (and were short of breath at rest), liver disease, or blindness; (10) changed residences during certain months of the year; (11) planned to move in the near future; or their HbA1c obtained at baseline was < 7.5%.

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Study Completion 2002-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah L. Krein, PhD RN, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI; Alan J. Pawlow, MD, Principal Investigator — John D. Dingell VA Medical Center, Detroit, MI; Rodney A. Hayward, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

REFERENCES:
- [Result] Krein SL, Vijan S, Choe HM, Hayward RA. Quality improvement strategies for type 2 diabetes. JAMA. 2006 Dec 13;296(22):2680; author reply 2681. doi: 10.1001/jama.296.22.2680-a. No abstract available. PMID 17164452
- [Result] Krein SL, Hofer TP, Kerr EA, Hayward RA. Whom should we profile? Examining diabetes care practice variation among primary care providers, provider groups, and health care facilities. Health Serv Res. 2002 Oct;37(5):1159-80. doi: 10.1111/1475-6773.01102. PMID 12479491
- [Result] Krein SL, Klamerus ML, Vijan S, Lee JL, Fitzgerald JT, Pawlow A, Reeves P, Hayward RA. Case management for patients with poorly controlled diabetes: a randomized trial. Am J Med. 2004 Jun 1;116(11):732-9. doi: 10.1016/j.amjmed.2003.11.028. PMID 15144909